CLINICAL TRIAL: NCT00626977
Title: Labor Analgesia With Ropivacaine Added to Clonidine. A Randomized Clinical Trial
Brief Title: Labor Analgesia With Ropivacaine and Clonidine
Acronym: LA
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Faculdade de Medicina de Botucatu, UNESP, Botucatu, Brasil (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Yara Marcondes Machado Castiglia, MD PhD, UPECLIN HC FM Botucatu Unesp
Other Study IDs: upeclin/HC/FMB-Unesp-07
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2008-02

CONDITIONS: Labor Pain
Keywords: Analgesia; Obstetrical; Anesthesia; Epidural; Newborn; Anesthetics, local; Clonidine; Pregnant women; Infant, newborn
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Ropivacaine; Clonidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- R: R group:15 mL of 0.125% ropivacaine (18.75 mg)
  Interventions: Drug: ropivacaine
- RC: RC group:0.0625% ropivacaine (9.375 mg) plus 75 ug clonidine
  Interventions: Drug: ropivacaine and clonidine

INTERVENTIONS:
Drug: ropivacaine — 15 ml of ropivacaine 0.125% peridural once
  Groups: R
Drug: ropivacaine and clonidine — 15 ml of ropivacaine 0.0625% plus 75 mcg clonidine
  Groups: RC

SUMMARY:
The aim of the present study was to examine, for pain relief during labor, the efficacy of two pharmacological approaches - the 0.125% ropivacaine alone and the 0.0625% ropivacaine added to 75 ug clonidine, both by epidural administration. The effect of the drugs on mother and newborn was also determined.

ELIGIBILITY:
Inclusion Criteria:

* Singleton healthy
* Full-term pregnancy
* American Society of Anesthesiologists physical status I or II

Exclusion Criteria:

* Patients who had received opioids
* History of hypersensitivity to local anesthetic or to clonidine
* Fetus showed signs of possible intrauterine suffering
* Fetus showed signs of possible neurological deficit

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women having requested epidural analgesia for labor and hers newborns
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2000-05; Primary Completion 2000-05 (Actual); Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giane Nakamura, MD PHd, Principal Investigator — College Study of Medicine
Locations (1):
- College of Medicine of Botucatu, Botucatu, São Paulo, Brazil

REFERENCES:
- [Derived] Nakamura G, Ganem EM, Modolo NS, Rugolo LM, Castiglia YM. Labor analgesia with ropivacaine added to clonidine: a randomized clinical trial. Sao Paulo Med J. 2008 Mar 6;126(2):102-6. doi: 10.1590/s1516-31802008000200007. PMID 18553032